CLINICAL TRIAL: NCT02667665
Title: Verification Study and Reactivity Study for the Validity of a Novel Dementia Rating Scale "QUick QUestion Scale" for Alzheimer's Disease Dementia
Brief Title: Verification Study and Reactivity Study for the Validity of QuQu Scale
Acronym: QuQu
Status: Completed | Type: Observational
Sponsor: Translational Research Center for Medical Innovation, Kobe, Hyogo, Japan (Other)
Collaborators: Daiichi Sankyo Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: TRIAD1412
Record Dates: First submitted 2016-01-26; First posted 2016-01-29 (Estimated); Last update posted 2017-06-02 (Actual); Status verified 2017-06

CONDITIONS: Alzheimer's Disease Dementia; Cognitive Concern Without Dementia
Keywords: Alzheimer's Disease Dementia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Alzheimer's Disease Dementia
- non-Dementia

SUMMARY:
Examine the construct validity, the test-retest reliability, the concurrent validity with the standard dementia rating scales and the reactivity of a novel dementia rating scale "QuQu scale: QUick QUestion scale" final for the evaluation of patients with Alzheimer's Disease Dementia and Mild Cognitive Impairment.

ELIGIBILITY:
Inclusion Criteria:

1. Alzheimer's Disease Dementia and patients with cognitive concern without Dementia
2. Written Informed consent by each subject and/or a legal representative, and study informant. If the doctor decides that the patient has no trouble in understanding this study, the written informed consent of a legal representative may be exempted. If not, this study needs a written informed consent by a legal representative and the patient except the case where the consent is hardly obtained due to the progression of the disease.

Exclusion Criteria:

1. patients with other types of dementia (e.g. vascular dementia, Levy body dementia, frontotemporal dementia)
2. patients with other diseases which cause secondary dementia prior to Alzheimer's Disease Dementia
3. patients with other severe neurological disease or psychiatric disorder without Alzheimer's Disease Dementia
4. patients with other medical conditions where the investigators determine that it is inappropriate for the subject of this study (e.g. inappropriate for the evaluation of dementia rating scale)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with Alzheimer's Disease Dementia and Mild Cognitive Impairment
Sampling Method: Non-Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2016-02-19 (Actual); Primary Completion 2016-11-15 (Actual); Study Completion 2016-11-15 (Actual)

PRIMARY OUTCOMES:
QuQu scale candidate | 12 weeks
Mini-Mental State Examination (MMSE) | 12 weeks
NPI-Caregiver Distress. Scale(NPI-D) | 12 weeks
Disability Assessment for Dementia (DAD) | 12 weeks
Clinical Dementia Rating | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Yu Nakamura, Professor, Study Chair — Kagawa University School of Medicine
Locations (1):
- Kagawa University School of Medicine, Kitagun, Kagawa-ken, Japan